CLINICAL TRIAL: NCT00184054
Title: Phase II Trial of Arsenic Trioxide With Ascorbic Acid in the Treatment of Adult Non-APL Acute Myelogenous Leukemia
Brief Title: Trial of Arsenic Trioxide With Ascorbic Acid in the Treatment of Adult Non-Acute Promyelocytic Leukemia (APL) Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing studies
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-02-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Arsenic Trioxide; Ascorbic Acid

ARMS (1):
- Arsenic Trioxide (ATO) Plus Ascorbic acid (Experimental): Arsenic Trioxide (ATO) given at 0.25 mg/kg/day intravenously for 25 days over a 35-day period.
  Ascorbic Acid given at 1000 mg/day intravenously every other day that ATO is given
  Interventions: Drug: Arsenic Trioxide (ATO); Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Arsenic Trioxide (ATO) — Arsenic Trioxide .25 mg/kg/day
Drug: Ascorbic Acid — Ascorbic Acid 1000 mg every other day for 25 days
  Other Names: Vitamin C

SUMMARY:
This clinical research study is for patients with acute myelogenous leukemia (in short AML) that did not respond to previous treatment or unable to receive chemotherapy.

Arsenic has been used as a drug for many centuries. While arsenic containing drugs were used in the past for cancer treatments, the major use of arsenic in western countries has been for the treatment of uncommon tropical illnesses, such as sleeping sickness. Recently, some new information suggests that arsenic in a form called arsenic trioxide may also be useful to treat some cancers of the blood, such as leukemia, lymphoma and myeloma. Studies from China and the USA showed that patients with a type of blood cancer called acute promyelocytic leukemia, whose disease failed to respond to other treatments, responded very well to arsenic trioxide. Studies done in laboratories in the United States have shown that arsenic can kill AML cells growing in culture dishes.

Ascorbic acid (vitamin C), a natural supplement in our diet, has long been involved with cancer prevention. Laboratory tests have shown that although arsenic trioxide by itself can kill AML cells in the test tube, when vitamin C is added to arsenic trioxide in a test tube, the death of the leukemia cells increases significantly.

The purpose of this study is to find out if the combination of arsenic trioxide (Trisenox) and ascorbic acid is effective in the treatment of patients who have AML. The second purpose is to study how the two drugs affect cells in the laboratory. Samples from the blood and bone marrow (the part of the body that makes blood cells) will be collected, at specific times during treatment, in order to study them in the laboratory. By studying blood and marrow cells, researchers hope to learn the mechanisms by which the drugs work.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-APL AML (FAB subtypes M0 - M7 but excluding M3) confirmed by myeloperoxidase stain and/or flow cytometry.
* For patients of age 18 or older - only refractory or relapsed AML will be included. Refractory disease is defined as newly diagnosed patients who fulfill ONE of the following criteria:

  * Patient aged 60 years or younger, who have failed to achieve a complete remission after at least two cycles of front line induction chemotherapy.
  * Patients of any age who have AML, that is post myelodysplastic syndrome (MDS), who failed to achieve a complete remission after at least one cycle of front line induction chemotherapy.
  * Patients aged 60 years or older who failed to achieve a complete remission after at least one cycle of front line induction chemotherapy.
* Newly diagnosed patients aged 55 or older who will not receive intensive anti-leukemia chemotherapy can also be enrolled.
* Post-myelodysplasia AML and secondary AML are included.
* Stem cell transplantation failures are included.
* Karnofsky performance status greater or equal to 50%.
* Adequate renal function (creatinine < 1.5 x ULN or creatinine clearance > 60 ml/min) and hepatic function (transaminases < 2.5 x ULN, serum total bilirubin < 3 mg/dl).
* Females of childbearing potential must have a negative serum pregnancy test prior to enrollment on the study, and both women and men must use an effective birth control method while on the study.
* Signed consent.

Exclusion Criteria:

* Newly diagnosed patients older than age 55 who:

  * Refuse chemotherapy when their treating physician recommends standard anti-leukemia induction chemotherapy.
  * Have a Karnofsky performance status of greater or equal to 70%, aged < 75 years and has no prior myelodysplastic syndrome.
  * Have a risk/benefit ratio that gives their treating physician good reason for administration of standard anti-leukemia induction chemotherapy.
* Patients who have already been treated with arsenics.
* CML in blastic crisis.
* Patients with cardiopathies including recurrent supraventricular arrhythmia and any type of sustained ventricular arrhythmia or conduction block (A-V block grade II or III, LBBB).
* Patients with HIV.
* Pregnant or breastfeeding women.
* QT interval > 460 msec in the presence of serum potassium > 4.0 mEq/L and magnesium > 1.8 mg/dL.
* Pre-existing neurotoxicity/neuropathy of Grade 2 or greater according to the NCI Common Toxicity Criteria Version 2.
* History of preexisting neurological disorders (grade 3 or higher by the NCI Common Toxicity Criteria; in particular, seizure disorders).
* Patients with an underlying medical condition that could be aggravated by the treatment or life threatening disease unrelated to AML as evaluated by the enrolling physician.
* Patients with active second malignancy, excluding adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Inability or unwillingness to comply with the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-04; Primary Completion 2009-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Douer, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study opened in April 2002 and closed in May 2008. All subjects were seen at USC.
Pre-assignment Details: The study has no pre-assignment. All subjects were given the same treatment.
Groups:
- Arsenic Trioxide (ATO) Plus Ascorbic Acid: All subjects received ATO 0.25 mg/kg/day intravenously for 25 days over a 35-day period and Ascorbic Acid 1000 mg/day intravenously every other day that ATO is given
Period: Overall Study
Arm/Group | Arsenic Trioxide (ATO) Plus Ascorbic Acid
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis.
Arm/Group | Arsenic Trioxide (ATO) Plus Ascorbic Acid
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response (Complete Remissions (CR) and Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: Complete Remission (CR): ANC >=1000/mcl, Platelet count >=100,000/mcl, Bone marrow <5% blasts. Complete Remission with incomplete blood count recovery (CRi): Same as CR but ANC may be <1,000/mcl and/or platelet count <100,000/mcl. Patients who failed to achieve CR or CRi after two cycles were considered treatment failures. Patients who did not complete at least two cycles were not evaluated for response.
Time Frame: Up to 1 year
Population: All subjects who received at least 2 cycles of treatment as part of this study are included in the analysis of response.
Measure: Number; unit: participants
Arm/Group | Arsenic Trioxide (ATO) Plus Ascorbic Acid
Number analyzed (Participants) | 11
participants
  CR | 1
  CRi | 5
  Treatment Failure | 4
  Not Evaluable | 1

2. Secondary Outcome: Number of Participants With Severe (Grades 3-5) Adverse Events
Description: Patients who received any amount of ATO plus Ascorbic Acid are included in the safety analyses.
Time Frame: Days 1, 8, 15, 21, 28, 35 of each cycle and at end of treatment (30 days after last dose or start of new therapy)
Measure: Number; unit: Participants
Arm/Group | Arsenic Trioxide (ATO) Plus Ascorbic Acid
Number analyzed (Participants) | 11
Participants
  Anorexia | 1
  Alanine aminotransferase increased | 1
  Conjunctivitis infective | 2
  Differentiation syndrome | 1
  Electrocardiogram QT corrected interval prolonged | 1
  Neuropathy: sensory | 1
  Sepsis | 4

ADVERSE EVENTS:
Time Frame: Days 1, 8, 15, 21, 28, 35 of each cycle and at end of treatment (30 days after last dose or start of new therapy)
Arm/Group | Arsenic Trioxide (ATO) Plus Ascorbic Acid
Serious Adverse Events (participants affected / at risk) | 11/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (ATO) Plus Ascorbic Acid (N=11)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 2 (2)
Differentiation syndrome (General disorders) | 1 (1) — Shortness of breath with hypoxia responding to steroids during hyperleukocytosi
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Neuropathy sensory (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (ATO) Plus Ascorbic Acid (N=11)
Anorexia (Metabolism and nutrition disorders) | 2 (4)
Cellulitis - hand (Infections and infestations) | 1 (1)
Localized edema (General disorders) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Fatigue (General disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 5 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No